CLINICAL TRIAL: NCT07161700
Title: A 6-Week, Multicenter, Open-Label, Monotherapy, Extension Study of SPT-300 in Adults With Major Depressive Disorder, With or Without Anxious Distress
Brief Title: An Open-Label Extension Study to Evaluate the Safety and Tolerability of SPT-300 (GlyphAllo) in Participants With Major Depressive Disorder, With or Without Anxious Distress (BUOY-1 OLE Study)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Seaport Therapeutics (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPT-300-2024-204; 2025-522347-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD); Major Depressive Disorder With Anxious Distress
Keywords: Major Depressive Disorder; Depressive Disorder; Depression; Anxiety; Mood Disorders; SPT-300; LYT-300; GlyphAllo; Glyph Allopregnanolone; BUOY-1 OLE Study; Anxious Distress; Open Label Extension Study
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPT-300 (Experimental): Participants will receive SPT-300 capsules once daily for 42 days
  Interventions: Drug: SPT-300

INTERVENTIONS:
Drug: SPT-300 — A prodrug of allopregnanolone, a small molecule drug
  Other Names: LYT-300; GlyphAllo; Glyph Allopregnanolone

SUMMARY:
This is an open-label, monotherapy, extension study to evaluate the safety and tolerability of SPT-300 (GlyphAllo) in adults with major depressive disorder (MDD), with or without anxious distress.

ELIGIBILITY:
Inclusion Criteria:

* Participant who completed treatment in Study SPT-300-2024-203 (i.e., participant who competed Visit 8 [Day 42] of Study SPT-300-2024-203 [BUOY-1 Study]).
* Women of childbearing potential (WOCP) must not plan to become pregnant during the course of the study or be currently breastfeeding. WOCP must agree to use a highly effective form of contraception during participation in the study and for 30 days after receiving the last dose of study treatment.
* Participant is willing and able to refrain from the use of drugs of abuse.

Exclusion Criteria:

* Participants who, in the opinion of the Investigator, medical monitor, or Sponsor, should not participate in the study.
* Participants who, in the judgment of the Investigator, were noncompliant with trial procedures or with study treatment administration during the double-blind study (BUOY-1 Study).
* Female participants with a positive urine pregnancy test result. Female participants may be enrolled without a negative urine test if they are surgically sterile or at least 2 years post-menopause.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability assessments based on Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and validated clinical scales and procedures | Up to Day 49
  Adverse events (AEs) are monitored from Day 1 to 49. A TEAE is as any AE with an onset after first dose of study treatment up to Day 49. Clinically significant abnormalities in clinical laboratory evaluations, ECGs, vital signs, physical examinations and Columbia Suicide Severity Rating Scale (C-SSRS) will be reported as TEAEs.

CONTACTS AND LOCATIONS:
Overall Officials: David Walling, Ph.D., Principal Investigator — Collaborative Neuroscience Research - Garden Grove
Locations (20):
- United States (12):
  - Seaport Investigator Site, Chino, California
  - Seaport Investigator Site, Glendale, California
  - Seaport Investigator Site, West Palm Beach, Florida
  - Seaport Investigator Site, Atlanta, Georgia
  - Seaport Investigator Site, Decatur, Georgia
  - Seaport Investigator Site, Boston, Massachusetts
  - Seaport Investigator Site, St Louis, Missouri
  - Seaport Investigator Site, Brooklyn, New York
  - Seaport Investigator Site, New York, New York
  - Seaport Investigator Site, Staten Island, New York
  - Seaport Investigator Site, North Canton, Ohio
  - Seaport Investigator Site, Irving, Texas
- Bulgaria (2):
  - Seaport Investigator Site, Plovdiv
  - Seaport Investigator Site, Sofia
- Czechia (2):
  - Seaport Investigator Site, Brno
  - Seaport Investigator Site, Prague
- Poland (4):
  - Seaport Investigator Site, Bialystok
  - Seaport Investigator Site, Bydgoszcz
  - Seaport Investigator Site, Gdansk
  - Seaport Investigator Site, Poznan